CLINICAL TRIAL: NCT01492998
Title: Study of the Role of the Biliary Salts Nuclear Receptor FXR in Hepatitis C Virus Replication
Brief Title: Role of FXR in Hepatitis C Virus Replication
Acronym: GGST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008.501-02
Record Dates: First submitted 2010-09-23; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C virus; Biliary salts; Farnesoid X receptor; Guggulsterone
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — pregna-4,17-diene-3,16-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guggulsterone (Experimental): One arm of 15 chronically HCV genotype one infected patients
  Interventions: Other: guggulsterone, a natural FXR antagonist.

INTERVENTIONS:
Other: guggulsterone, a natural FXR antagonist. — Gugulipid®, natural extract from Commiphora mukul tree, containing 2.5% guggulsterone

SUMMARY:
In vitro in the hepatitis C virus (HCV) replicon system, modulation of the biliary salts nuclear receptor FXR by either agonists or antagonists respectively increases or decreases the replication of HCV (J Hepatol, 2008, 48: 192-9). One antagonist of FXR is a vegetal sterol, guggulsterone, that is extracted from the Commiphora mukul tree and that has already been given safely to hyper cholesterolemic patients in a clinical trial (JAMA 2003, 290: 765-72). The aim of this trial is to test the effect of the FXR antagonist guggulsterone given orally, three times a day, on the viral load in 15 HCV genotype 1 chronically infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients infected by HCV genotype 1, with anti-HCV antibodies, non responders to at least one first line of therapy
* Viral load > 1 x 105 UI/mL for more than 6 months and not treated for at least the last two months.
* METAVIR score < F4

Exclusion Criteria:

* Alcohol intake > 20 g/day
* Immuno - suppressive therapy
* Obesity BMI > 30, diabetes
* Dyslipidemia requiring specific therapy
* Liver cirrhosis or carcinoma
* HIV or HBV co-infections
* Other liver diseases
* Major organ failures
* Therapy with cytochrome P450 metabolized drugs

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Evolution of the HCV plasmatic viral load while taking the FXR inhibitor guggulsterone. | One week

SECONDARY OUTCOMES:
Modification of the fraction of the circulating viral forms associated with apolipoprotein B | One week

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trépo, MD, Prof., Principal Investigator — Hospices Civils de Lyon; Marianne Maynard, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Department of hepatology, Hospices Civils de Lyon, Hôtel Dieu, Lyon, France

REFERENCES:
- [Derived] Scholtes C, Andre P, Trepo C, Cornu C, Remontet L, Ecochard R, Bejan-Angoulvant T, Gueyffier F. Farnesoid X receptor targeting for hepatitis C: study protocol for a proof-of-concept trial. Therapie. 2012 Sep-Oct;67(5):423-7. doi: 10.2515/therapie/2012058. Epub 2012 Dec 18. PMID 23241251